CLINICAL TRIAL: NCT05842876
Title: Renal NIRS Monitoring to Detect Coarctation of the Aorta - A Pilot Study
Brief Title: Happy Baby Hearts Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1710; SMPH\PEDIATRICS\NEONATO (Other: UW Madison); Protocol Version 3/29/2024 (Other: UW Madison); A536757 (Other: UW Madison)
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Coarctation of Aorta
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Caregiver + Low Risk neonates: Participants in the nursery who are expected to be lower risk for CoA
  Interventions: Device: Continuous Renal NIRS Monitoring; Diagnostic Test: Standard Clinical Care; Other: Satisfaction Survey
- Caregiver + Medium to High Risk neonates: Participants in the NICU who are expected to be at a higher risk for CoA
  Interventions: Diagnostic Test: Standard Clinical Care
- Nurses in the Newborn Nursery: Nurses who work at the Meriter Hospital, Inc. Newborn Nursery
  Interventions: Other: Satisfaction Survey

INTERVENTIONS:
Device: Continuous Renal NIRS Monitoring — Renal oxygenation data collected every 6 seconds
  Groups: Caregiver + Low Risk neonates
Diagnostic Test: Standard Clinical Care — q6 h BP, q6 h Pulse ox, Echo at 24-72h
  Groups: Caregiver + Low Risk neonates
Diagnostic Test: Standard Clinical Care — Renal oxygenation data collected every 6 seconds, q6 h BP, continuous Pulse ox, Echo at 12-72h
  Groups: Caregiver + Medium to High Risk neonates
Other: Satisfaction Survey — Survey to assess which method of monitoring is preferred
  Groups: Caregiver + Low Risk neonates; Nurses in the Newborn Nursery

SUMMARY:
The goal of this observational study is to determine the feasibility of renal Near Infrared Spectroscopy (NIRS) monitoring in the newborn nursery for newborns at low risk of coarctation of the aorta (CoA). The main questions it aims to answer are:

* whether continuous renal NIRS monitoring is feasible;
* whether NIRS monitoring results in higher nursing and parent/caregiver satisfaction than current standard monitoring; and,
* whether participants who develop CoA will spend a smaller proportion of time within the normal range than patients who do not have CoA.

Participants will be observed through continuous renal oxygenation monitoring with NIRS.

ELIGIBILITY:
Neonate Inclusion Criteria:

* Delivered at ≥ 35 weeks of gestation
* <12 hours of age
* Inpatient at Meriter Hospital, Inc. NICU or Newborn Nursery or AFCH PICU or NICU
* Diagnosed as at risk for CoA

Neonate Exclusion Criteria:

* Major congenital anomalies of the kidney
* Attending physician's discretion to not place sensors due to clinical concerns
* In the researcher's medical opinion, there is a significant likelihood that the neonate would not survive the first 3 days of life

Primary Caregiver Inclusion Criteria:

* Able to understand and the willing to sign a written informed consent document
* Willing to comply with all study procedures and be available for the duration of the study
* Birth parent (i.e., the parent who gave birth to the baby) who is the primary caregiver of a neonate who is eligible to participate in study
* Agrees to enroll neonate into study
* Aged 15 years or older
* Pregnant mother with a baby diagnosed prenatally as at risk for CoA will be eligible for the study. They must also meet the following criteria:
* Require an "arch watch care plan" as a results of prenatal ultrasonography findings
* Agree to enroll offspring into the study at birth

Primary Caregiver Exclusion Criteria:

* Subject is unable to provide informed consent, including subjects who are in foster care and subjects within state custody
* Pregnant woman who does not plan to maintain custody of the child after birth, such as instances of adoption or surrogacy

Newborn Nursery Nursing Staff:

* All Newborn Nursery nursing staff at Meriter Hospital, Inc.'s Newborn Nursery are eligible to participate

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Neonates admitted to the nursery or NICU at Meriter Hospital, Inc. or UWHealth Kids - American Family Children's Hospital (AFCH) who are ≥ 35 weeks' gestation and have a prenatally identified concern for coarctation of the aorta.
  2. Primary parent/guardian of neonate.
  3. Nursing staff at Meriter Hospital, Inc.'s Newborn Nursery
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Percent of time monitored | Up to 2 weeks post-delivery, on average
  Amount of time continuously monitored will be calculated
Count of adverse and unexpected events | Up to 2 weeks post-delivery
  All adverse and unexpected events will be recorded

SECONDARY OUTCOMES:
Change in nursing satisfaction with renal NIRS monitoring | Study start to one year later
  A subjective description of survey responses in addition to determining which method of monitoring is preferred: NIRS vs. Enhanced BP/Pulse ox checks. Survey will be conducted at the beginning of the study, and one year later.
Parent/caregiver satisfaction with renal NIRS monitoring | Up to 2 weeks post-delivery, on average
  A subjective description of survey responses in addition to determining which method of monitoring is preferred: NIRS vs. Enhanced BP/Pulse ox checks
Renal oxygen trends | Through study completion, approximately 1 year
  A permutation test will be used to compare the distribution of proportions (of time spent within normal range) between the two groups (CoA vs. normal)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin, Madison, Wisconsin
  - Meriter Hospital, Inc., Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh Y. Evaluation of a child with suspected congenital heart disease. Paediatrics and Child Health 2018, 28(12): 556-561
- [Background] Levey A, Glickstein JS, Kleinman CS, Levasseur SM, Chen J, Gersony WM, Williams IA. The impact of prenatal diagnosis of complex congenital heart disease on neonatal outcomes. Pediatr Cardiol. 2010 Jul;31(5):587-97. doi: 10.1007/s00246-010-9648-2. Epub 2010 Feb 18. PMID 20165844
- [Background] Gomez-Montes E, Herraiz Garcia I, Escribano Abad D, Rodriguez Calvo J, Villalain Gonzalez C, Galindo Izquierdo A. Application of a Global Multiparameter Scoring System for the Prenatal Prediction of Coarctation of the Aorta. J Clin Med. 2021 Aug 20;10(16):3690. doi: 10.3390/jcm10163690. PMID 34441986
- [Background] Maskatia SA, Kwiatkowski D, Bhombal S, Davis AS, McElhinney DB, Tacy TA, Algaze C, Blumenfeld Y, Quirin A, Punn R. A Fetal Risk Stratification Pathway for Neonatal Aortic Coarctation Reduces Medical Exposure. J Pediatr. 2021 Oct;237:102-108.e3. doi: 10.1016/j.jpeds.2021.06.047. Epub 2021 Jun 26. PMID 34181988
- [Background] Korcek P, Stranak Z, Sirc J, Naulaers G. The role of near-infrared spectroscopy monitoring in preterm infants. J Perinatol. 2017 Oct;37(10):1070-1077. doi: 10.1038/jp.2017.60. Epub 2017 May 4. PMID 28471443
- [Background] Hazle MA, Gajarski RJ, Aiyagari R, Yu S, Abraham A, Donohue J, Blatt NB. Urinary biomarkers and renal near-infrared spectroscopy predict intensive care unit outcomes after cardiac surgery in infants younger than 6 months of age. J Thorac Cardiovasc Surg. 2013 Oct;146(4):861-867.e1. doi: 10.1016/j.jtcvs.2012.12.012. Epub 2013 Jan 12. PMID 23317940